CLINICAL TRIAL: NCT00124098
Title: An Open-Label Study of Aranesp® (Darbepoetin Alfa) Administration Once Every Four Weeks in Anaemic Chronic Kidney Disease (CKD) Subjects
Brief Title: An Evaluation of Aranesp® in Subjects With Anaemic Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030112
Record Dates: First submitted 2005-06-30; First posted 2005-07-27 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Kidney Disease
Keywords: Chronic Kidney Disease (CKD); anemia, clinical trial; darbepoetin alfa; Aranesp®; Amgen
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp® (darbepoetin alfa)

SUMMARY:
The purpose of this study is to assess if Aranesp® administered once every 4 weeks to chronic kidney disease subjects is safe and efficacious in maintaining haemoglobin levels greater than or equal to 100 g/L.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic kidney disease and not expected to initiate dialysis for the duration of the study
* Creatinine clearance greater than 15 and less than 40 mL/min as estimated by the Cockroft-Gault equation:

  * Creatinine Clearance = (140-age in years) x body weight in kg/serum creatinine (mg/dL) x 72.
  * For women, the value will be multiplied by 0.85
* Receiving stable every other week subcutaneous doses of Aranesp®.
* A stable dose is defined as less than or equal to 25% change in Aranesp® dose over the 6-week period immediately prior to enrollment and with no more than

  1 missed dose over this period
* At least two haemoglobin values within the target range of 100 to 130 g/L obtained at least 1 week apart and within 5 weeks of the baseline visit
* Subjects must have a haemoglobin of 100 to 130 g/L at eligibility/baseline
* Serum ferritin greater than or equal to 100 mg/L or transferrin saturation greater than or equal to 19.5%
* Serum vitamin B12 and folate levels must be above the lower limit of the normal range of the local laboratory
* Before any study specific procedure is performed, the subject must provide informed consent for participation in the study

Exclusion Criteria:

* Anticipating, scheduled for, or a prior recipient of a kidney transplant
* Uncontrolled hypertension (blood pressure greater than 160/100 mmHg during the eligibility/baseline period on 2 separate measurements)
* Congestive heart failure (New York Heart Association [NYHA] class III or IV)
* Clinical evidence of severe hyperparathyroidism (parathyroid hormone level greater than 1500 pg/mL or biopsy-proven bone marrow fibrosis)
* Major surgery within 12 weeks before enrollment (excluding vascular access surgery)
* Active chronic inflammatory process
* Currently receiving antibiotic therapy for systemic infection
* ALT or AST greater than 2 times the upper limit of normal range
* Known positive HIV antibody or positive hepatitis B surface antigen
* Clinical evidence of current malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia
* Red blood cell transfusions within 8 weeks before eligibility visit or active bleeding
* Systemic hematologic disease (e.g., sickle cell anaemia, myelodysplastic syndromes, hematologic malignancy, myeloma, haemolytic anaemia)
* Psychiatric or any other disorder which may impact (in the judgment of the Investigator) the ability to give informed consent for participation in this study
* Pregnant or breast feeding women
* All subjects must practice adequate contraception in the judgment of the Investigator, during the course of their participation in the trial
* Previous entry in this study
* Treatment with an investigational agent other than Aranesp® or device within 30 days before the first dose of study drug or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Haemoglobin level

SECONDARY OUTCOMES:
Aranesp® doses
Adverse events
Laboratory parameters
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Disney A, Jersey PD, Kirkland G, Mantha M, Charlesworth JA, Gallagher M, Harris D, Gock H, Mangos GJ, Macmillan J, Liu W, Viswalingam A. Darbepoetin alfa administered monthly maintains haemoglobin concentrations in patients with chronic kidney disease not receiving dialysis: a multicentre, open-label, Australian study. Nephrology (Carlton). 2007 Feb;12(1):95-101. doi: 10.1111/j.1440-1797.2006.00757.x. PMID 17295668
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20030112.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/